CLINICAL TRIAL: NCT03886532
Title: GI Medical Cannabis Registry and Pharmacology
Brief Title: GI Medical Cannabis Study on IBD
Acronym: GIMEDCAN
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding/support
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 18-015221
Record Dates: First submitted 2019-01-14; First posted 2019-03-22 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases; Neuropathic Pain
MeSH Terms: conditions — Inflammatory Bowel Diseases; Neuralgia | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — We will consent subjects to retain microsampling samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Medical Marijuana: Those subject taking only medical marijuana as standard of care. Will collect registry data and collect blood samples.
  Interventions: Other: Medical Marijuana
- CBD only products: Those subjects taking only CBD products as standard of care. Will collect registry data and collect blood samples.
  Interventions: Other: Medical Marijuana

INTERVENTIONS:
Other: Medical Marijuana — registry and blood samples

SUMMARY:
Create a registry that will described the natural history and landscape of medical cannabis product use in patients with chronic abdominal pain or inflammatory bowel disease.

Quantitatively describe the pharmacokinetic (PK) profile of select medical cannabis products in patients with chronic neuropathic (abdominal) pain or inflammatory bowel disease.

To create an educational program for families that have participated in the research for those families who opt for this component. Although these are not research in nature, they are a direct result of the proposed research and are included in the protocol to demonstrate the study's deliverables.

DETAILED DESCRIPTION:
Although the state-level legalization of cannabis for medical use allows access for patients, its use closely resembles the dietary supplement market. In 1994, the Dietary Supplement Health and Education Act (DSHEA) was passed, allowing dietary supplements to be available to consumers without prior proof of quality, safety, or efficacy. The goal of the legislation was to allow consumer access to potentially beneficial therapies without the delay from research and regulatory body approval. Unfortunately, the research did not follow, and now the dietary supplement market is an unregulated industry that is fraught with fraudulent claims and unsafe, contaminated, and/or adulterated products, many of which have unknowingly harmed individuals. Similar to dietary supplements, cannabis as a therapy is largely unstudied, with over 100 active constituents, each of which has its own potential pharmacologic actions. Different blends of these constituents have the potential to reap significant therapeutic benefits. Unfortunately, the traditional drug development paradigm has not been performed for these products.

Objectives:

The overall goal of this research is to characterize the current use and disposition of medical cannabis including cannabidiol (CBD) products being administered to children and adults as standard of care, and to understand the pharmacokinetics (PK) and pharmacodynamics (PD) of compounds in these medical cannabis products. An additional component of this study is to provide educational feedback to families and care providers to provide evidenced-based dosing guidance for these products to patients with qualifying gastrointestinal disorders.

1. The primary objective is to describe the natural history and landscape of medical cannabis including CBD use in patients with qualifying gastrointestinal disorders, specifically chronic abdominal pain and inflammatory bowel disease. There will be a specific focus on the variability of products and routes of administration.
2. The secondary objective is to quantitatively describe the PK profile of select medical cannabis products in patients with these gastrointestinal disorders.
3. Another secondary objective is to create an educational program for families that have participated in the research, for those families who opt for this component.

Study Design:

This is a prospective observational cohort study.

Setting/Participants:

Persons who are receiving medical cannabis as therapy, who have a diagnosis of chronic abdominal pain or inflammatory bowel disease.

Study Interventions and Measures:

1. Investigators will collect demographics, data regarding utilization, formulation, indications, and concomitant medications. Investigators will do an initial intake and perform follow-up to inquire about any changes in medications or medical history on a monthly basis.
2. Once four subjects have been recruited who are taking the same formulation of a cannabis product, the study team will contact them for consent for the PK portion of the study. Investigators will collect five samples with a microsampling technique. If at any point there is a change in symptoms and/or product, Investigators will collect another five samples. The purpose of the collection is to assay for cannabis-related compounds [(e.g. Tetrahydrocannabinol (THC), CBD)] to quantitatively describe the PK profile.
3. Educational sessions will be created for research subjects and families who opt to participate. Investigators will hold meetings which may be in person or online and invite those interested participants to learn about our findings. This will be done at approximately six-month intervals throughout the study, or when it is deemed appropriate by the study team to share than information.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who consume cannabis products in a state which has legalized medical cannabis for the treatment of inflammatory bowel disease and chronic neuropathic (abdominal) pain.
2. Individuals who have a diagnosis of Inflammatory Bowel Disease or chronic neuropathic (abdominal) pain.

Exclusion Criteria:

1. Consumption of cannabis products that are not obtained from a state-sanctioned dispensary.
2. Non English speaking individuals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed with inflammatory bowel disease (IBD) and are taking medical marijuana or cannabidiol (CBD) legally
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms | 1 year
  Relief of primary indication (perceived therapeutic benefit of product) reported via parent or caregiver on a 1-10 Lichert scale with 1 being minimally effective and 10 being extremely effective.

SECONDARY OUTCOMES:
Patient or caregiver reported side effects | 1 year
  There is no particular scale or instrument being used to collect this data. Patients and caregivers are reporting on any perceived side effects from the medication.
Changes in drug concentrations | 1 year
  To assess changes in pharmacokinetic levels in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Athena F Zuppa, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia

IPD SHARING:
Plan to Share IPD: No